CLINICAL TRIAL: NCT05977530
Title: Teaching Young Children Swim Survival Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Schwebel, University Professor of Psychology & Associate Vice President for Research Facilities & Infrastructure, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300011508
Record Dates: First submitted 2023-07-18; First posted 2023-08-04 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Drowning
MeSH Terms: conditions — Drowning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- self-rescue training (Experimental): children will receive self-rescue training from a certified instructor
  Interventions: Behavioral: self-rescue training

INTERVENTIONS:
Behavioral: self-rescue training — children will receive training for self-rescue if they are alone in water

SUMMARY:
This study is designed to evaluate whether commercially-available swim self-rescue schools are effective to teach children ages 12-23 months to stay safely alive floating in the water (or grasping the pool's edge) without adult intervention. The investigators will measure children's water self-rescue skills at baseline and then they will engage in commercially-available training over the course of several weeks. The investigators will then measure their skills again. Assessments will be conducted using a standardized protocol with a certified lifeguard present. Parents will also complete a short survey concerning child and family demographics and child and family swim and lifeguard training experience.

ELIGIBILITY:
Inclusion Criteria:

* child ages 12-23 months
* enrolled in self-rescue course at participating swim facility

Exclusion Criteria:

* medical conditions counter-indicating training in water
* previous experience in self-rescue swim courses

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Youth Safety Lab, University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data with qualified researchers upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after all primary results are published. They will remain available for at least 3 years.
Access Criteria: Contact Study PI David Schwebel.

REFERENCES:
- [Derived] Schwebel DC, Johnston A. Toddler drowning prevention through self-rescue: can 1-year-old children learn to float? Inj Prev. 2025 Nov 11:ip-2025-045688. doi: 10.1136/ip-2025-045688. Online ahead of print. PMID 41219144

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Self-rescue Training
Started | 50
Completed | 48
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — injury unrelated to research participation. Unable to enter swimming pool to participate in protocol | 1

BASELINE CHARACTERISTICS:
Population: children ages 12-23 months
Arm/Group | Self-rescue Training
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.45 (0.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 43
  More than one race | 4
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Children's Self-rescue Ability
Description: Assessment of whether children demonstrates ability to engage independently and safely in water, without adult assistance. This was measured through a standardized behavioral observation of children's behavior in a swimming pool. It was scored in a binary fashion as "yes" or "no", with each child in the study scored either "yes" or "no".
Time Frame: at completion of training intervention program, an anticipated average of 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Self-rescue Training
Number analyzed (Participants) | 48
Participants | 48
Statistical Analysis 1: Comparison: Self-rescue Training; Test type: Superiority; p < .01, Wilcoxon (Mann-Whitney); comparison of ranks in Wilcoxon = 0

ADVERSE EVENTS:
Time Frame: About 5 minutes at baseline assessment and about 10 minutes during post-intervention assessment at week 4
Description: Does not differ from clinicaltrials.gov definitions.
Arm/Group | Self-rescue Training
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT05977530/Prot_SAP_000.pdf